CLINICAL TRIAL: NCT00953160
Title: Pilot Study to Evaluate the Cutera RF Device for Reduction in Size of Localized Areas of the Body, Including, But Not Limited to, Areas on the Abdomen, Leg, and Arm
Brief Title: Radio Frequency (RF) Device for Reduction in Size of Localized Areas of the Body
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The preliminary data from this pilot study did not indicate efficacy.
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-09-TF-02
Record Dates: First submitted 2009-08-04; First posted 2009-08-06 (Estimated); Results first posted 2011-03-17 (Estimated); Last update posted 2023-09-18 (Actual); Status verified 2023-08

CONDITIONS: Cellulite
Keywords: Cellulite; Adipose tissue; Circumference; Reduction; Thigh; Abdomen; Flank
MeSH Terms: conditions — Cellulite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RF treatment (Experimental): Abdomen, flank or thigh treated with RF device
  Interventions: Device: Cutera Radio Frequency Device

INTERVENTIONS:
Device: Cutera Radio Frequency Device — Up to three treatments, one pass, dosage range of 15-60 kJ.
  Other Names: Callisto, TruForm, TruSculpt

SUMMARY:
The purpose of this study is to evaluate the Cutera radio frequency (RF) device for the new indication of reduction in size of localized areas of the body.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the Cutera radio frequency device for the new indication of reduction in size of localized areas of the body, including, but not limited to, areas on the abdomen, leg, and arm.

At investigator's discretion, each subject will receive up to three treatments and will be scheduled for two follow-up visits after the final treatment. The treated area will be measured and photographed ar each visit for analysis. Subjects will also be weighted at each visit and asked to fill out a survey during follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Female or Male
* Minimum age of 18 years
* Non-smoking for at least 3 months and willing to refrain from smoking for the duration of the study.
* Post-menopausal, or on birth control with no plans to become pregnant for the duration of the study (female only)
* Minimum Body Mass Index of 20
* Visible fat in the area to be treated Area to be treated to measure at least 20.0mm in vertical fold, as measured with industry standard fat caliper
* Subject must be able to read, understand and sign the Consent Form
* Subject must adhere to the follow-up schedule and study instructions
* Subject must adhere to the same diet and/or exercise routine throughout the study, and agree to maintain the same weight throughout the study (within 6 lbs of initial weight)

Exclusion Criteria:

* Significant weight fluctuation (+/-10 lbs) in the past 6 months
* Taking weight-loss medications/supplements
* Participation in any other clinical study
* Cellulite treatment within 3 months of the treatment
* Surgical or non-surgical treatments to the target area in the last 12 months, e.g., liposuction
* Prior treatment to the target area within the last 12 months
* Arteriosclerosis or weakened blood vessels
* Heart disease
* Thromboembolic disease
* Diagnosed or documented immune system disorders
* Bleeding disorders.
* Presence of uncontrolled hypertension
* Taking prescription anticoagulants
* History of keloid formation
* Malignant tumors in the target area
* Diabetes
* Any disease or condition that could impair wound healing
* Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, scars, large moles
* Infection in the target area
* Implanted electrical device(s)
* Pregnant or lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2009-04; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Biesman, MD, Principal Investigator; Jacqueline Calkin, MD, Principal Investigator; Stephen Ronan, MD, Principal Investigator; Scott Kramer, MD, Principal Investigator; Adele Makow, MD, Principal Investigator; Barry DiBernardo, MD, Principal Investigator
Locations (5):
- United States (5):
  - Blackhawk Plastic Surgery, Danville, California
  - Renu LaserSpa, Dublin, California
  - Calkin/Boudreaux Dermatology Associates, Sacramento, California
  - New Jersey Plastic Surgery, Montclair, New Jersey
  - Nashville Center for Laser and Facial Surgery, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study subjects were recruited in the medical clinic 01/01/09 through 01/13/10.
Groups:
- Radiofrequency (RF) Treatment: Abdomen, flank or thigh treated with RF device (average of 2 treatments and average dosage of 30kJ)
Period: Overall Study
Arm/Group | Radiofrequency (RF) Treatment
Started | 76
Completed | 49
Not Completed | 27
Not completed — Lost to Follow-up | 23
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Radiofrequency (RF) Treatment
Number analyzed (Participants) | 76
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 76
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 76

OUTCOME MEASURES:

1. Primary Outcome: Change in Circumference (cm)
Time Frame: Baseline and 6 months post final treatment
Measure: Mean (Standard Deviation); unit: Centimeters (cm)
Arm/Group | Radiofrequency (RF) Treatment
Number analyzed (Participants) | 49
Centimeters (cm)
  Abdomen | -0.5 (2.2)
  Thigh | 0.6 (4.7)
  Flank | -1.4 (2.1)

2. Secondary Outcome: Subject Satisfaction
Time Frame: Baseline and 6 months post final treatment
Arm/Group | Radiofrequency (RF) Treatment
Number analyzed (Participants) | 0

3. Secondary Outcome: The Number of Participants With Adverse Events
Description: At each visit (treatment and follow-up) or until resolution of AEs
Time Frame: Up to 6 months after the last treatment
Measure: Number; unit: Participants
Arm/Group | Radiofrequency (RF) Treatment
Number analyzed (Participants) | 49
Participants
  Edema | 1
  Lumps | 3

ADVERSE EVENTS:
Time Frame: 6 months
Description: Subjects were assessed and followed up for adverse events at 6 weeks, 3 months and 6 months after the RF treatment.
Arm/Group | Radiofrequency (RF) Treatment
Serious Adverse Events (participants affected / at risk) | 0/49
Other Adverse Events (participants affected / at risk) | 3/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Radiofrequency (RF) Treatment (N=49)
Lumps (Injury, poisoning and procedural complications) | 3 (49)

LIMITATIONS AND CAVEATS:
Early termination of the study resulting in analysis of small numbers of subjects, and technical issues with repeatability and reproducibility of circumference measurements leading to termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
"The Doctor will not publish or present the results of the Study, or speak publicly about it, unless Cutera has first had a reasonable opportunity to review and comment on the contents of the proposed presentation or publication."